CLINICAL TRIAL: NCT03988621
Title: Improving Self-Care of Informal Caregivers of Adults With Heart Failure
Brief Title: Improving Self-care of Heart Failure Caregivers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Barbara Riegel, PHD, RN, Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01NR018196 (NIH)
Record Dates: First submitted 2019-05-22; First posted 2019-06-17 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Self-care; Self-efficacy; Heart Failure; Stress; Support Systems
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The study was based on the Transactional Model of Stress and Coping. Stressful experiences such as caregiving demand - circumstances that give rise to real or perceived stress - are construed as person-environment transactions. Primary appraisal of demand involves assessment of its significance, which results in perceived burden. Secondary appraisal involves assessment of the resources available to cope with it. These appraisals lead to the coping effort. Without successful coping, self-care is poor, which decreases health status in caregivers. The virtual support intervention [ViCCY ("Vicky") - Virtual Caregiver Coach for You] addressed both appraisal and coping.
Who Masked: Investigator
Masking Description: The investigator was blinded to the assignment of participant to the two different arms in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Caregivers randomized to the intervention ViCCY received 10 sessions of virtual health coaching by trained health coaches over 6 months with content based on the theoretical framework (the Transactional Model of Stress and Coping) and prior research. In addition, they received the same health information as that provided to the caregivers in the control arm. Sessions were provided through tablets. We helped caregivers gain the knowledge and skills needed to achieve self-identified health goals through self-care using motivational interviewing. We focused on identifying personal values, solving problems, and transforming goals into action. ViCCY was standardized in a treatment manual. Because stress does not affect all people equally, the intervention was tailored to individual appraisals and the factors most likely to influence demand and perceived burden.
  Interventions: Behavioral: ViCCY
- Control (No Intervention): The control group received Health Information (HI) delivered through the internet.

INTERVENTIONS:
Behavioral: ViCCY — Virtual Caregiver Coach for You
  Arms: Intervention

SUMMARY:
Informal caregiving is demanding and stressful. Caregivers of adults with heart failure (HF) report significant stress and poor self-care. Health coaching, a support intervention, may relieve stress and promote self-care in HF caregivers. Few studies have tested the cost-effectiveness of support interventions for caregivers. Even less is known about the effect of caregiver support interventions on HF outcomes. We developed and tested a virtual support intervention (ViCCY ("Vicky")-Virtual Caregiver Coach for you), in HF caregivers. Using randomized controlled trial (RCT) design, we enrolled informal HF caregivers with poor self-care (Health Self-Care Neglect scale score>=2), randomizing them 1:1 to an intervention or control group. Both groups received Health Information (HI) delivered through the Internet, but the ViCCY caregiver group also received 10 health coaching support sessions tailored to individual issues. The control group had access to the same HI resources over the same interval, using the same Internet program, but without coaching support. At baseline and 3, 6, 9, and 12 months, we collected self-reported data on self-care, stress, coping, and health status. At 6 months, we compared ViCCY to HI alone to assess intervention efficacy using intent-to-treat analysis. A sample of 250 caregivers (125/arm) was enrolled to provide >90% power to detect significant differences between the groups on the primary outcome of self-care (Aim 1). We collected quality adjusted life years (QALYs) and health care resource use in caregivers over 12 months to assess cost-effectiveness of ViCCY (Aim 2). To explore the effect of caregiver outcomes on HF patients' outcomes (hospitalization rates, hospital days, mortality rates, QALYs) over a 12-month period (Aim 3) and knowing that not all HF patients would enroll, we consented a subgroup of 93 HF patients cared for by these caregivers to explore the effect of caregiver self-care on patient outcomes. If shown to be efficacious and cost-effective, our virtual health coaching intervention can easily scaled to support millions of caregivers worldwide. This application addresses the NINR strategic plan and is directly responsive to PA-18-150.

DETAILED DESCRIPTION:
We used a randomized controlled trial (RCT) design, randomizing informal heart failure (HF) caregivers meeting our inclusion and exclusion criteria 1:1 to an intervention or control group. After collecting baseline data, we block randomized the caregivers to achieve equal distribution of key variables in each condition. We will block randomize on caregiver sex (male/female), relationship to patient (e.g., spouse), and race. Sex and relationship are factors known to influence perceived caregiving burden and receptivity to intervention. Race was included to assure group balance. The randomization sequence was generated a priori by a statistician independent of the study investigators using a randomly permuted blocks algorithm to ensure equal distribution of these variables in each study arm. The Project Manager notified study staff and participants of their group assignment (intervention or control) by telephone, email or message, as preferred by the individual. Investigators and all staff involved in collecting assessment data were blinded to group assignment until after the data were locked. The health coach providing the intervention and the caregiver participants were not be blinded. All baseline data were collected prior to randomizing. Timing of follow-up assessments were based on day of randomization.

The study intervention was provided to individual caregivers. All caregivers (both groups) were provided with access to an Internet site with excellent health information (HI). The virtual support intervention (ViCCY ["Vicky"] - Virtual Caregiver Coach for You) was provided through tablet devices provided to caregivers in the intervention group. We provided tablets to all the caregivers, assuring that they had wireless network access so they can access the Internet site providing HI content. Caregivers in the control group received only HI but caregivers in the intervention group received 10 sessions of ViCCY over 6 months.

ELIGIBILITY:
Inclusion Criteria: Informal caregiver of adults with heart failure providing care at least 8 hours/week, reporting poor self-care on screening (Health Self-Care Neglect scale score >=2 based on our pilot data), able to complete the protocol, e.g., adequate vision and hearing, and English speaking were required for enrollment.

Exclusion Criteria: Cognitive impairment (Telephone Interview for Cognitive Status [TICS] <25), Participation in another clinical trial of a support intervention, Untreated major psychiatric illness (Use of anti-anxiety/antidepressant medicines was acceptable and will be adjusted in analysis if group imbalance is identified).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Hospital Heart and Vascular Clinic, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share the data internally with doctoral students and post-doctoral trainees instead of sharing the data widely with external sources. Internal sharing will allow our trainees to complete meaningful studies using secondary analysis techniques and to finish their programs in a timely fashion. When all our analyses have been completed we will share the data through a public source.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication of our major trial data, we will share data with Penn trainees.
Access Criteria: The Principal Investigator will personally review requests from students for use of the data. She will approve requests based on the importance of the questions asked. She will personally oversee progress in analysis and the publication of abstracts and articles based on the data.

REFERENCES:
- [Result] Riegel B, Quinn R, Hirschman KB, Thomas G, Ashare R, Stawnychy MA, Bowles KH, Aryal S, Wald JW. Health Coaching Improves Outcomes of Informal Caregivers of Adults With Chronic Heart Failure: A Randomized Controlled Trial. Circ Heart Fail. 2024 Jul;17(7):e011475. doi: 10.1161/CIRCHEARTFAILURE.123.011475. Epub 2024 Jun 21. PMID 38904103
- [Derived] Riegel B, Quinn R, Hirschman KB. A longitudinal comparative analysis of sustained benefit of a self-care intervention for caregivers of adults with heart failure. BMC Nurs. 2025 Nov 22;24(1):1501. doi: 10.1186/s12912-025-04123-4. PMID 41272616

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 677 caregivers were screened for eligibility from a regional HF referral center in the US from August 2019- November 2022. 502 were eligible, 50% of those declined participation and 26% did not meet inclusion criteria.
  250 caregivers were enrolled and consented for participation. 93 patients associated with the enrolled caregivers were consented to participate. Patient enrollment exceeded the targeted goal of 40.
Pre-assignment Details: Enrolled caregivers were stratified by race, relationship to caregiver, and sex prior to assignment of intervention arm.
Groups:
- Intervention: Caregivers randomized to the intervention (Virtual Caregiver Coach for You [ViCCY]) received 10 sessions of virtual health coaching by health coaches over 6 months. Intervention content was based on the theoretical framework (Transactional Model of Stress and Coping) and prior research. Sessions were individual and virtual (provided using tablets). The health coaches helped caregivers gain the knowledge and skills needed to achieve their self-identified health goals through self-care. We focused on identifying personal values, solving problems, and transforming goals into action. ViCCY is standardized in a treatment manual. Because stress does not affect all people equally, the intervention was tailored to individual appraisals and the factors most likely to influence demand and perceived burden.
  ViCCY: Virtual Caregiver Coach for You
- Control: Caregivers in the control group received Health Information delivered through a Samsung tablet programmed with health information websites. They were asked to spend at least 30 minutes weekly using the computer tablet provided to them by the study team to access the recommended websites
Period: Overall Study
Arm/Group | Intervention | Control
Started (Caregivers) | 167 | 176
Started (Caregivers) | 125 | 125
3-Month Survey(Caregivers) | 93 | 103
6-Month Survey(Caregivers) (Primary study endpoint at 6 months.) | 93 | 101
9-Month Survey(Caregivers) (Some participants who did not complete data at 6 months were available again at 9- and 12-months. But, the primary analysis was done with 6-month data.) | 103 | 104
12-Month Survey(Caregivers) | 95 | 101
Started (Patients) | 42 | 51
12 Month Survey/Completed(Patients) (Patient primary study endpoint at 12 months.) | 26 | 31
Completed (Caregivers and Patients: 12 Month Timepoint Complete) | 121 | 132
Not Completed | 46 | 44
Not completed — Lost to Follow-up | 16 | 17
Not completed — Withdrawal by Subject | 14 | 7
Not completed — Patient Lost to Follow Up | 15 | 15
Not completed — Patient death | 1 | 5

BASELINE CHARACTERISTICS:
Population: This was a study of caregivers so the population studied reflects the 250 caregivers enrolled. In addition, as an exploratory aim, we enrolled a sample of 93 patients. The analysis of patient data was not the focus of this study so that Participant Flow focuses on caregivers.
Groups:
- Intervention: Caregivers randomized to the intervention (Virtual Caregiver Coach for You [ViCCY]) received 10 sessions of virtual health coaching by health coaches over 6 months. Intervention content was based on the theoretical framework (Transactional Model of Stress and Coping) and prior research. Sessions were individual and virtual (provided using tablets). The health coaches helped caregivers gain the knowledge and skills needed to achieve their self-identified health goals through self-care. We focused on identifying personal values, solving problems, and transforming goals into action. ViCCY is standardized in a treatment manual. Because stress does not affect all people equally, the intervention was tailored to individual appraisals and the factors most likely to influence demand and perceived burden.
  ViCCY: Virtual Health Coaching for You
- Control: Caregivers randomized to the control group received Health Information on Samsung tablets. They were asked to spend at least 30 minutes weekly using the computer tablets to access recommended websites.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 167 | 176 | 343
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age is measured in years. Population: Analysis population consists of 250 caregivers and 93 patients.
  Years
    Caregiver Age: number analyzed (Participants) | 125 | 125 | 250
    Caregiver Age | 55.4 (13.78) | 55.3 (13.55) | 55.3 (13.64)
    Patient Age: number analyzed (Participants) | 42 | 51 | 93
    Patient Age | 56.1 (16.34) | 56.9 (15.37) | 56.5 (15.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Self-reported sex Population: Analysis population consists of 250 caregivers and 93 patients
  Participants
    Caregiver Data: number analyzed (Participants) | 125 | 125 | 250
    Caregiver Data: Female | 106 | 107 | 213
    Caregiver Data: Male | 19 | 18 | 37
    Patient Data: number analyzed (Participants) | 42 | 51 | 93
    Patient Data: Female | 10 | 10 | 20
    Patient Data: Male | 32 | 41 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported ethnicity (Hispanic vs. not Hispanic) Population: Analysis population consists of 250 caregivers and 93 patients
  Participants
    Caregiver Data: number analyzed (Participants) | 125 | 125 | 250
    Caregiver Data: Hispanic or Latino | 5 | 4 | 9
    Caregiver Data: Not Hispanic or Latino | 119 | 120 | 239
    Caregiver Data: Unknown or Not Reported | 1 | 1 | 2
    Patient Data: number analyzed (Participants) | 42 | 51 | 93
    Patient Data: Hispanic or Latino | 1 | 0 | 1
    Patient Data: Not Hispanic or Latino | 41 | 50 | 91
    Patient Data: Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported information collected at baseline. Population: Analysis population consists of 250 caregivers and 93 patients
  Participants
    Caregiver Data: number analyzed (Participants) | 125 | 125 | 250
    Caregiver Data: American Indian or Alaska Native | 0 | 0 | 0
    Caregiver Data: Asian | 1 | 3 | 4
    Caregiver Data: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregiver Data: Black or African American | 35 | 39 | 74
    Caregiver Data: White | 79 | 76 | 155
    Caregiver Data: More than one race | 6 | 5 | 11
    Caregiver Data: Unknown or Not Reported | 4 | 2 | 6
    Patient Data: number analyzed (Participants) | 42 | 51 | 93
    Patient Data: American Indian or Alaska Native | 0 | 1 | 1
    Patient Data: Asian | 0 | 0 | 0
    Patient Data: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Patient Data: Black or African American | 8 | 12 | 20
    Patient Data: White | 31 | 37 | 68
    Patient Data: More than one race | 2 | 0 | 2
    Patient Data: Unknown or Not Reported | 1 | 0 | 1
Self Care Maintenance [Mean (Standard Deviation); unit: units on a scale] — Self-Care Maintenance is one scale of the Self-Care Inventory. This scale measures efforts to maintain one's health through health promoting practices. Scores range from 0-100. Higher scores indicate better self-care. The focus of this intervention and analysis was on Self-Care Maintenance. The composite reliability coefficient was 0.73 and the global reliability index for multidimensional scales was 0.85. Test-retest reliability was 0.81 after 10 days in 125 volunteers drawn from a US sample. This theoretically derived instrument has construct validity. Population: 250 caregivers analyzed. One caregiver did not provide sufficient data for the Self Care Inventory survey and thus has a missing value for the score.
  units on a scale
    number analyzed (Participants) | 124 | 125 | 249
    (all) | 68.8 (16.1) | 68.2 (15.7) | 68.5 (15.9)
Years as caregiver [Median (Inter-Quartile Range); unit: years] — Years spent caregiving were self-reported by caregivers at baseline. Population: 250 caregivers analyzed. One caregiver did not provide sufficient data for the Years Caregiving survey question and thus has a missing value for the score.
  years
    number analyzed (Participants) | 124 | 125 | 249
    (all) | 3.75 [1.1 to 9.2] | 3.00 [1.6 to 8] | 3.25 [1.3 to 8.7]
Hours caregiver per day [Mean (Standard Deviation); unit: Hours] — Hours typically spent daily in caregiving were self-reported at baseline by caregivers. Specifically, caregivers were prompted to report "How many hours per day do you care for him or her? (hours/day)" Population: 250 caregivers analyzed. Three caregivers did not provide sufficient data for this measure at baseline.
  Hours
    number analyzed (Participants) | 123 | 124 | 247
    (all) | 8.2 (7.5) | 7.9 (7.5) | 8.1 (7.5)
Health Self-care Neglect (HSCN) scale [Mean (Standard Deviation); unit: units on a scale] — The Health Self-Care Neglect Scale measures specific behaviors that the caregiver self-reports as neglecting. Scores range from 0-9 with higher scores indicating more self-neglect. In testing recently conducted with baseline data, reliability was assessed with composite reliability model-based estimates. Concurrent validity was assessed by correlating the HSCN scale total score with the maintenance scale score of the Self-Care Inventory. Population: 250 Caregivers Analyzed
  units on a scale
    number analyzed (Participants) | 125 | 125 | 250
    (all) | 4.9 (2.1) | 5.0 (2.1) | 4.9 (2.1)
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — The Perceived Stress Scale measures how stressful an individual perceives their life to be. This scale contains 14 questions, and respondents rate themselves on a scale of 0 (never) to 4 (very often) for each question. Scores range from 0-56. Higher scores indicate higher perceived stress. Population: 250 caregivers analyzed. Two caregivers did not provide sufficient data for this measure at baseline.
  units on a scale
    number analyzed (Participants) | 123 | 125 | 248
    (all) | 25.9 (7.5) | 26.5 (7.7) | 26.2 (7.6)
Active Coping Subscale [Mean (Standard Deviation); unit: units on a scale] — The Ways of Coping Scale measures coping processes and identifies the thoughts and actions used to cope when facing a specific stressful encounter. The scale has three subscales used in this study (active, minimization, and avoidance coping). Items are rated 0 (not used) to 3 (used a great deal). This active coping subscale has 15 items and scores that range from 0 - 45. Higher scores indicate more use of active methods to cope with stress. It is reliable (alpha 0.95) and has construct validity. This instrument has been used numerous times in studies with older adult caregivers. Population: 250 caregivers analyzed. Six caregivers did not provide sufficient data for this measure at baseline.
  units on a scale
    number analyzed (Participants) | 120 | 124 | 244
    (all) | 22.6 (9.1) | 22.9 (10.3) | 22.7 (9.7)
Avoidance Coping Subscale [Mean (Standard Deviation); unit: units on a scale] — The Ways of Coping Scale measures coping processes and identifies the thoughts and actions used to cope when facing a specific stressful encounter. The scale has three subscales used in this study (active, minimization, and avoidance coping). Items are rated 0 (not used) to 3 (used a great deal). This avoidance coping subscale has 10 items and scores that range from 0 - 30. Higher scores indicate more use of avoidance methods such as wishful thinking to cope with stress. It is reliable (alpha 0.95) and has construct validity. Population: 250 caregivers analyzed. Five caregivers did not provide sufficient data for this measure at baseline.
  units on a scale
    number analyzed (Participants) | 120 | 125 | 245
    (all) | 9.0 (5.9) | 10.7 (6.4) | 9.9 (6.2)
Minimization Coping Subscale [Mean (Standard Deviation); unit: units on a scale] — The Ways of Coping Scale measures an individual's coping processes and identifies the thoughts and actions an individual used to cope when facing a specific stressful encounter. The scale has three subscales used in this study (active, minimization, and avoidance coping). Items are rated 0 (not used) to 3 (used a great deal). This subscale measuring minimization coping has 10 items and scores that range from 0 - 30. Higher scores indicate that the person uses minimization methods (efforts to detach from the unpleasant situation) to cope with stress. Population: 250 caregivers analyzed. Eight caregivers did not provide sufficient data for this measure at baseline.
  units on a scale
    number analyzed (Participants) | 119 | 123 | 242
    (all) | 11.8 (5.4) | 12.9 (5.6) | 12.3 (5.5)
Short Form (SF)-36 Physical Health Status [Mean (Standard Deviation); unit: units on a scale] — The SF-36 measures overall health status along 8 domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. The scale uses both Likert-scale questions and yes or no questions. Scores can be summed as physical and mental health. Physical health is calculated using items reflecting physical functioning, physical role and bodily pain. Scores are standardized 0-100 with higher scores indicating better physical functioning. Population: 250 caregivers analyzed. Seven caregivers did not provide sufficient data for this measure at baseline.
  units on a scale
    number analyzed (Participants) | 120 | 123 | 243
    (all) | 48.0 (10.1) | 47.3 (9.6) | 47.6 (9.8)
Short Form (SF)-36- Mental Health Status [Mean (Standard Deviation); unit: units on a scale] — The SF-36 measures overall health status along 8 domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. The scale uses both Likert-scale questions and yes or no questions. Scores can be summed as physical and mental health. Mental health is calculated using items reflecting mental health, emotional role functioning, and social functioning. Scores are standardized 0-100 with higher scores indicating better mental functioning. Population: 250 caregivers analyzed. Seven caregivers did not provide sufficient data for this measure at baseline.
  units on a scale
    number analyzed (Participants) | 120 | 123 | 243
    (all) | 43.2 (12.3) | 41.1 (12.2) | 42.1 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Health Self-Care Neglect (HSCN) Scale
Description: The Health Self-Care Neglect (HSCN) scale measures an individual's neglect of self-care behaviors. It consists of 9 yes or no questions. Scores range from 0-9. Higher scores indicating more self-care neglect.
Time Frame: The primary outcome was analyzed at 6 months (baseline compared to 6 months) but data were collected at 9- and 12-months to assess sustainability.
Population: Number of participants analyzed differs across timepoints due to participant attrition, missing data due to nonresponse, and/or missed study timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: Caregivers randomized to the intervention received 10 sessions of virtual health coaching by trained health coaches over 6 months. Content of the sessions was guided by the Transactional Model of Stress and Coping and prior research. Sessions were provided virtually using tablets. We called the intervention ViCCY (virtual caregiver coach for you) and sought to help caregivers gain the knowledge and skills needed to achieve their health goals through self-care. We focus on identifying personal values, solving problems, and transforming goals into action. ViCCY is standardized in a treatment manual. Because stress does not affect all people equally, the intervention is tailored to individual appraisals and the factors most likely to influence demand and perceived burden.
  ViCCY: Virtual Health Coaching for You
- Control: The control group received only Health Information (HI) delivered through the internet.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 125
score on a scale
  HSCN Baseline Score | 4.89 (2.07) | 4.97 (2.12)
  HSCN 3 Month Score: number analyzed (Participants) | 93 | 103
  HSCN 3 Month Score | 3.09 (2.07) | 3.50 (2.17)
  HSCN 6 Month Score: number analyzed (Participants) | 93 | 100
  HSCN 6 Month Score | 2.67 (2.09) | 3.49 (2.16)
  HSCN 9 Month Score: number analyzed (Participants) | 97 | 99
  HSCN 9 Month Score | 2.34 (1.99) | 3.02 (2.24)
  HSCN 12 Month Score: number analyzed (Participants) | 95 | 100
  HSCN 12 Month Score | 2.57 (2.10) | 3.09 (2.17)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.04, Mixed Models Analysis — The p-value for the group-by-time interaction is presented, as well as the estimated mean and confidence interval for difference in 6-month change between intervention and treatment groups; Mean Difference (Net) = -0.65, 95% CI 2-sided [-1.27 to -0.03] — Mean HSCN scale scores of participants in the intervention group were estimated to decrease by 0.65 (95% CI: -1.27 to -0.03) units more than that of participants in the control group from baseline to 6-months

2. Primary Outcome: Change in the Self-Care Inventory, Maintenance Scale
Description: The Self-Care Inventory is a 20 item inventory with 3 embedded scales (self-care maintenance, monitoring, and management). The outcome used in this study was the 8-item Self-Care Maintenance Scale. Responses are added and standardized to range from 0-100. A higher score indicates better self-care.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention: Caregivers randomized to the ViCCY intervention
  ViCCY: Virtual Health Coaching for You
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 125
score on a scale
  Self Care Maintenance, Baseline Score: number analyzed (Participants) | 124 | 125
  Self Care Maintenance, Baseline Score | 68.83 (16.09) | 68.15 (15.73)
  Self Care Maintenance, 6 Month Score: number analyzed (Participants) | 92 | 100
  Self Care Maintenance, 6 Month Score | 79.86 (12.29) | 72.85 (12.35)
  Self Care Maintenance, 12 Month Score: number analyzed (Participants) | 95 | 101
  Self Care Maintenance, 12 Month Score | 76.62 (13.26) | 74.58 (14.61)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.01, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 5.05, 95% CI 2-sided [1.12 to 8.98] — Mean Self Care Inventory scale scores of participants in the intervention group were estimated to increase by 5.05 (95% CI: 1.12 to 8.98) units more than that of participants in the control group from baseline to 6-months

3. Secondary Outcome: Change in the Perceived Stress Scale (PSS)
Description: The Perceived Stress Scale (PSS), a 14-item instrument that provides a global rating of an individual's belief in the severity and frequency of stressful experiences during the last month. The Perceived Stress Scale includes 14 items designed to assess symptoms of stress and global measures of the degree of stress experienced in the past month. Each item is scored from 0 (never) to 4 (very often), with total sum scores ranging from 0 to 56; higher scores indicate higher perceived stress. In prior test, Cronbach's alpha of the scale ranged from 0.84 to 0.86, and was 0.91 for older African American and European American females.
Time Frame: Main analysis was Baseline to 6 months. Data will be analyzed at 12 months to determine sustainability of intervention effect.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Intervention: Caregivers randomized to the intervention ViCCY (Virtual Health Coaching for You).
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 125
Score on a scale
  PSS Baseline Score: number analyzed (Participants) | 123 | 125
  PSS Baseline Score | 25.91 (7.48) | 26.49 (7.73)
  PSS 6 Month Score: number analyzed (Participants) | 92 | 100
  PSS 6 Month Score | 19.73 (6.97) | 25.20 (8.71)
  PSS 12 Month Score: number analyzed (Participants) | 94 | 101
  PSS 12 Month Score | 20.76 (8.39) | 24.00 (9.02)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -4.50, 95% CI 2-sided [-6.48 to -2.52] — Mean PSS scale scores of participants in the intervention group were estimated to decrease by 4.50 (95% CI: -6.48 to -2.52) units more than that of participants in the control group from baseline to 6-months

4. Secondary Outcome: Change in the Ways of Coping Questionnaire
Description: We used a 30-item modification of the original 42-item questionnaire developed by Lazarus in 1985. We measured these coping styles: active, avoidance, and minimization. The instrument uses a 4-point Likert-scale response format (0 = not used to 3 = used a great deal). Scores range from 0-45, 0-30, and 0-30 for the active, avoidance and minimization subscales, respectively. Higher scores indicate greater use of particular coping styles.
Time Frame: The primary analysis was at 6 months (baseline compared to 6 months) but data were collected at 9- and 12-months to assess sustainability.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Intervention: Caregivers randomized to the intervention ViCCY (Virtual Caregiver Coach for You)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 125
Score on a scale
  Avoidance Coping Baseline Score: number analyzed (Participants) | 120 | 125
  Avoidance Coping Baseline Score | 9.04 (5.86) | 10.72 (6.37)
  Avoidance Coping 3 Month Score: number analyzed (Participants) | 90 | 101
  Avoidance Coping 3 Month Score | 8.95 (5.72) | 9.01 (6.22)
  Avoidance Coping 6 Month Score: number analyzed (Participants) | 91 | 98
  Avoidance Coping 6 Month Score | 8.82 (5.86) | 11.85 (6.18)
  Avoidance Coping 9 Month Score: number analyzed (Participants) | 96 | 99
  Avoidance Coping 9 Month Score | 9.84 (5.73) | 10.89 (6.83)
  Avoidance Coping 12 Month Score: number analyzed (Participants) | 92 | 100
  Avoidance Coping 12 Month Score | 8.61 (6.32) | 10.54 (6.10)
  Active Coping Baseline Score: number analyzed (Participants) | 120 | 124
  Active Coping Baseline Score | 22.56 (9.14) | 22.92 (10.29)
  Active Coping 3 Month Score: number analyzed (Participants) | 91 | 100
  Active Coping 3 Month Score | 24.88 (8.95) | 21.52 (10.06)
  Active Coping 6 Month Score: number analyzed (Participants) | 90 | 98
  Active Coping 6 Month Score | 27.36 (9.54) | 25.50 (10.66)
  Active Coping 9 Month Score: number analyzed (Participants) | 96 | 99
  Active Coping 9 Month Score | 27.99 (8.71) | 27.55 (9.09)
  Active Coping 12 Month Score: number analyzed (Participants) | 92 | 98
  Active Coping 12 Month Score | 26.31 (9.59) | 26.00 (10.43)
  Minimize Coping Baseline Score: number analyzed (Participants) | 119 | 123
  Minimize Coping Baseline Score | 11.78 (5.39) | 12.89 (5.64)
  Minimize Coping 3 Month Score: number analyzed (Participants) | 91 | 102
  Minimize Coping 3 Month Score | 11.91 (5.29) | 11.99 (5.79)
  Minimize Coping 6 Month Score: number analyzed (Participants) | 92 | 98
  Minimize Coping 6 Month Score | 12.16 (4.36) | 13.87 (5.66)
  Minimize Coping 9 Month Score: number analyzed (Participants) | 96 | 99
  Minimize Coping 9 Month Score | 11.95 (4.58) | 12.15 (4.73)
  Minimize Coping 12 Month Score: number analyzed (Participants) | 92 | 100
  Minimize Coping 12 Month Score | 12.03 (5.14) | 13.18 (5.98)
Statistical Analysis 1: Comparison: Intervention vs Control; Active Coping Subscale; Test type: Superiority; p = 0.099, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 2.16, 95% CI 2-sided [-0.41 to 4.73]
Statistical Analysis 2: Comparison: Intervention vs Control; Avoidance Coping Subscale; Test type: Superiority; p = 0.25, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -0.88, 95% CI 2-sided [-2.38 to 0.62] — Estimated difference may not be consistent with difference sample means presented in outcome measure data table
Statistical Analysis 3: Comparison: Intervention vs Control; Minimization Coping Subscale; Test type: Superiority — The p-value for the group-by-time interaction is presented, as well as the estimated mean and confidence interval for difference in 6-month change between intervention and treatment groups; p = 0.68, Mixed Models Analysis; Mean Difference (Net) = -0.31, 95% CI 2-sided [-1.81 to 1.18]

5. Secondary Outcome: Change in Health Status as Measured by the Short Form-36 (Physical and Mental Health Status)
Description: Medical Outcomes Study Short Form (SF-36): measure of physical and mental health.The SF-36 has 36 items formatted in scales of varied format (3-, 5- and 6-pt scales and dichotomous [yes/no] scales). Each component score is standardized a 0-100 point scale. Higher values represent better health status. Reliability is varied samples is typically 0.80. Convergent and divergent validity have been demonstrated in various populations, including caregivers. A benefit of using the SF-36 is that it is one of the common data elements.
Time Frame: Main analysis Baseline to 6 months. Sustainability assessed at 12 months.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Intervention: Caregivers randomized to the intervention ViCCY (Virtual Caregiving Coaching for You)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 125 | 125
Score on a scale
  SF36 Physical Component Baseline Score: number analyzed (Participants) | 120 | 123
  SF36 Physical Component Baseline Score | 48.02 (10.11) | 47.25 (9.57)
  SF36 Physical Component 6 Month Score: number analyzed (Participants) | 92 | 99
  SF36 Physical Component 6 Month Score | 47.84 (9.84) | 48.18 (9.52)
  SF36 Physical Component 12 Month Score: number analyzed (Participants) | 94 | 101
  SF36 Physical Component 12 Month Score | 49.10 (9.33) | 47.57 (10.95)
  SF36 Mental Component Baseline Score: number analyzed (Participants) | 120 | 123
  SF36 Mental Component Baseline Score | 43.17 (12.27) | 41.06 (12.21)
  SF36 Mental Component 6 Month Score: number analyzed (Participants) | 92 | 99
  SF36 Mental Component 6 Month Score | 48.18 (10.43) | 42.73 (12.10)
  SF36 Mental Component 12 Month Score: number analyzed (Participants) | 94 | 101
  SF36 Mental Component 12 Month Score | 46.87 (11.27) | 44.33 (11.78)
Statistical Analysis 1: Comparison: Intervention vs Control; Physical Health Score; Test type: Superiority; p = 0.27, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -1.32, 95% CI 2-sided [-3.68 to 1.04]
Statistical Analysis 2: Comparison: Intervention vs Control; Mental Health Score; Test type: Superiority; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 3.35, 95% CI 2-sided [0.17 to 6.53] — Mean Mental Health scores of participants in the intervention group were estimated to increase by 3.35 (95% CI: 0.17 to 6.53) units more than that of participants in the control group from baseline to 6-months

6. Secondary Outcome: Change in the Caregivers' SF-6D (Short Form Six-dimension) Scores
Description: The SF-6D uses preference weights derived from the SF-36. The Short-Form Six-Dimension (SF-6D) provides a way to use the SF-36 in economic evaluation by estimating a preference-based single index measure for health from these data using general population values. The SF-6D score represents caregiver quality of life at a given timepoint. Higher SF-6D Scores are better.
Time Frame: Measured at baseline, 3, 6, 9, and 12 months; primary analysis baseline to 12 months
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Control: Caregivers in the control group received Health Information (HI) delivered through the internet.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 81 | 85
Score on a scale
  Baseline SF-6D | 0.696 (0.105) | 0.675 (0.132)
  6 Month SF-6D | 0.733 (0.119) | 0.688 (0.128)
  12 Month SF-6D | 0.731 (0.107) | 0.690 (0.116)

7. Secondary Outcome: Difference in Caregivers' Hospital and Provider Events
Description: Healthcare resource use was self-reported by caregivers when they were telephoned at each follow-up period, asking about utilization since the last interview date. The self-reported healthcare use comprised 5 major categories: hospitalizations, emergency department (ED) visits, diagnostic and therapeutic procedures, ambulance services, and home care services. A bottom-up cost account approach was used, wherein the sum of resources times their unit price yielded the total costs associated with healthcare resource use. Unit prices were measured using the 2021 Medical Expenditure Panel Survey (MEPS) (https://meps.ahrq.gov/mepsweb), an annual survey on the financing and use of medical care in the United States collected by the Agency for Healthcare Research and Quality (AHRQ).
Time Frame: Data were collected at Baseline, 3, 6, 9, and 12 months. The primary analysis was done using the baseline to 12 month period.
Population: At 12-months we had 209 caregivers available for the analysis; 15 were missing healthcare utilization data. We excluded 1 outlier who was in the hospital a long time. Then we had 193 in the final sample. Some of the 193 caregivers included in the analysis skipped one or two or even more follow-up interviews. However, caregivers were asked to report their healthcare utilization since the last follow-up and thus these records were able to be included in analysis.
Measure: Mean (Standard Deviation); unit: Dollars
Groups:
- Intervention: Caregivers randomized to the intervention ViCCY (Virtual Caregiving Coach for You)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 93 | 100
Dollars
  Healthcare Cost 0-1 Month: number analyzed (Participants) | 92 | 93
  Healthcare Cost 0-1 Month | 59.703 (281.566) | 67.004 (379.774)
  Healthcare Cost 0-3 Month: number analyzed (Participants) | 93 | 96
  Healthcare Cost 0-3 Month | 247.539 (1223.542) | 955.193 (4262.877)
  Healthcare Cost 0-6 Month: number analyzed (Participants) | 93 | 98
  Healthcare Cost 0-6 Month | 1155.871 (2577.653) | 1585.167 (5448.238)
  Healthcare Cost 0-9 Month: number analyzed (Participants) | 93 | 99
  Healthcare Cost 0-9 Month | 1347.139 (3018.211) | 2007.453 (6889.446)
  Healthcare Cost 0-12 Month | 1811.245 (3228.807) | 3121.488 (8123.811)

8. Other Pre Specified Outcome: Difference in Patient Hospitalization Rate
Description: For the 93 patients enrolled, the medical record was reviewed to capture hospitalization count. The aim was to explore the effect of caregiver outcomes (self-care) on HF patient outcomes. We hypothesize that at 12 months, HF patients whose caregivers improve vs. not improve in self-care (regardless of treatment group) will have Lower hospitalization rates. A comparison of patients' hospitalization counts which occurred between 6 and 12 month timepoints was conducted between those caregivers who exhibited a self care improvement from baseline to 6 month timepoint and those caregivers who did not exhibit a self care improvement from the baseline to 6 month timepoint.
Time Frame: Count of patient hospitalizations that occurred between 6 and 12 months (following the intervention, which ended at 6 months)
Population: The study sample includes 93 patients total. Because analysis focuses on patient outcomes during months 6 to 12 of the study, 4 patients were excluded from analysis of patient health outcomes due to death occurring between baseline and 6-month study timepoint. Among the remaining 89 enrolled patients, 15 did not provide sufficient data to determine whether self care improved from baseline to six months. Thus, a sample of 74 patients was analyzed.
Measure: Mean (Standard Deviation); unit: Hospitalization Count
Groups:
- Enrolled Patients With Caregivers Who Improved in Self Care: Enrolled patients with caregivers who exhibited improvement in self care from baseline to 6 months.
- Enrolled Patients With Caregivers Who Did Not Improve in Self Care: Enrolled patients with caregivers who did not exhibit improvement in self care from baseline to 6 months.
Arm/Group | Enrolled Patients With Caregivers Who Improved in Self Care | Enrolled Patients With Caregivers Who Did Not Improve in Self Care
Number analyzed (Participants) | 48 | 26
Hospitalization Count | 0.40 (0.89) | 0.31 (0.62)
Statistical Analysis 1: Comparison: Enrolled Patients With Caregivers Who Improved in Self Care vs Enrolled Patients With Caregivers Who Did Not Improve in Self Care; Test type: Superiority; p = 0.5433, Regression, zero inflated poisson; Mean Difference (Final Values) = 1.3472, 95% CI 2-sided [0.5153 to 3.5218] — Estimation accounts for the zero-inflated distribution of hospitalization count, thus estimate is inconsistent with mean values in the Outcome Measure Data table

9. Other Pre Specified Outcome: Patient Hospitalization Days
Description: For the 93 patients enrolled, the medical record was reviewed to capture hospitalization days. The aim was to explore the effect of caregiver outcomes (self-care, stress, coping, health status) on HF patient outcomes. We hypothesize that at 12 months, HF patients whose caregivers improve vs. not improve in self-care (regardless of treatment group) will have Lower hospitalization rates. A comparison of patients' hospitalization days which occurred between 6 and 12 month timepoints was conducted between those caregivers who exhibited a self care improvement from baseline to 6 month timepoint and those caregivers who did not exhibit a self care improvement from the baseline to 6 month timepoint.
Time Frame: Count of patient hospitalization days which occurred between 6 and 12 month timepoints
Population: The study sample includes 93 patients total. Because analysis focuses on patient outcomes during months 6 to 12 of the study, 4 patients were excluded from analysis of patient health outcomes due to death occurring between baseline and six month study timepoint. Among the remaining 89 enrolled patients, 15 did not provide sufficient self care data from baseline to six months. Lastly, one outlier was excluded with 148 hospital days in 6 months.A sample of 73 patients was analyzed.
Measure: Mean (Standard Deviation); unit: hospitalization days count
Groups:
- Patients of Caregivers Who Exhibited Improvement in Self Care: Patients of Caregivers who exhibited improvement in self care from baseline to 6 months.
- Patients of Caregivers Who Did Not Exhibit Improvement in Self Care: Patients of Caregivers who did not exhibit improvement in self care from baseline to 6 months.
Arm/Group | Patients of Caregivers Who Exhibited Improvement in Self Care | Patients of Caregivers Who Did Not Exhibit Improvement in Self Care
Number analyzed (Participants) | 48 | 25
hospitalization days count | 3.85 (8.71) | 3.04 (12.16)
Statistical Analysis 1: Comparison: Patients of Caregivers Who Exhibited Improvement in Self Care vs Patients of Caregivers Who Did Not Exhibit Improvement in Self Care; Test type: Superiority; p = 0.9173, Zero-inflated poisson regression; Mean Difference (Final Values) = 1.0143, 95% CI 2-sided [0.7766 to 1.3247]

10. Other Pre Specified Outcome: Patient Mortality Rates
Description: For the 93 patients enrolled, the medical record was reviewed to measure mortality. The aim was to explore the effect of caregiver outcomes (self-care, stress, coping, health status) on HF patient outcomes. We hypothesize that at 12 months, HF patients whose caregivers improve vs. not improve in self-care (regardless of treatment group) would have lower mortality rates. A comparison of patient mortality occurring between 6 and 12 months was conducted between those caregivers who improved in self care during the intervention period (baseline to 6 months) and those caregivers who did not improve in self care.
Time Frame: Patient mortality occurring between months 6-12 of the study (following the intervention period)
Population: The study sample includes 93 patients total. Because analysis focuses on patient outcomes during months 6 to 12 of the study, 4 patients were excluded from analysis of patient health outcomes due to death occurring between baseline and six month study timepoint. Among the remaining 89 enrolled patients, 15 did not provide sufficient data to determine whether self care improved from baseline to six months. Thus, a sample of 74 patients was analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients of Caregivers Who Exhibited Improvement in Self Care | Patients of Caregivers Who Did Not Exhibit Improvement in Self Care
Number analyzed (Participants) | 48 | 26
Participants
  Alive | 47 | 26
  Dead | 1 | 0
Statistical Analysis 1: Comparison: Patients of Caregivers Who Exhibited Improvement in Self Care vs Patients of Caregivers Who Did Not Exhibit Improvement in Self Care; Test type: Superiority; p = 0.6486, Fisher Exact

11. Other Pre Specified Outcome: Change in the Patients' Quality Adjusted Life Years (QALYs) Measured With the SF-6D (Short Form Six-dimension) Derived From the Short Form-36
Description: This measure of quality adjusted life years (QALY) is derived from the SF-36. It was used in the cost-effectiveness analysis. The SF-6D uses preference weights derived from the SF-36. The Short-Form Six-Dimension (SF-6D) provides a way to use the SF-36 in economic evaluation by estimating a preference-based single index measure for health from these data using general population values. The SF-6D score represents patient quality of life at a given timepoint, while the QALY represents the area under the curve of patient quality of life from baseline to 12-month timepoints. A QALY value of one equates to one year in perfect health. Higher quality adjusted life years (QALYs) are better.
Time Frame: QALYs were measured at baseline, 3, 6, 9, and 12 months. But this analysis focused on the baseline to 12 month period.
Population: 49 patients provided complete SF36 data at both baseline and 12 month timepoints.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Enrolled Patients With Caregivers Who Exhibited Improvement in Self Care: Enrolled patients with caregivers who improved in self care from baseline to 6 months.
- Enrolled Patients With Caregivers Who Did Not Improve in Self Care: Enrolled patients with caregivers who did not improve in self care from baseline to 6 months.
Arm/Group | Enrolled Patients With Caregivers Who Exhibited Improvement in Self Care | Enrolled Patients With Caregivers Who Did Not Improve in Self Care
Number analyzed (Participants) | 33 | 16
Score on a scale | 0.67 (0.11) | 0.68 (0.1)
Statistical Analysis 1: Comparison: Enrolled Patients With Caregivers Who Exhibited Improvement in Self Care vs Enrolled Patients With Caregivers Who Did Not Improve in Self Care; Test type: Superiority; p = 0.6791, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrolled caregivers at baseline, 3-month, 6-month, 9-month, and 12-month study timepoints.
Description: Caregiver and patient adverse event data was provided by caregivers at each study timepoint (baseline, 3-month, 6-month, 9-month, and 12-month). Caregiver self-reporting of adverse event information was verified against chart reviews performed at the 12-month. Adverse events not reported by the caregiver but discovered during chart reviews were also recorded for the caregiver and the patient.
Groups:
- Intervention: Caregivers randomized to the intervention ViCCY will receive 10 front-loaded sessions of virtual health coaching by trained registered nurses over 6 months with content based on the theoretical framework (based on the Transactional Model of Stress and Coping) and prior research. Sessions are provided using Samsung tablets that are also programmed with health information.
  For the primary aim it was hypothesized that 6 months after enrollment. the caregivers, randomized to receive the intervention would have more improvement in self-care, greater reductions in stress, greater improvement in coping and greater improvements in health status measured as the Sf. 3, 6, mental and physical component scores.
- Health Information: The caregivers got augmented standard care with health information programmed on on Samsung tablets
- Intervention (Patient): The study also aims to explore the effect of caregiver outcomes on patient outcomes. The hypothesis is that if the caregiver is less stressed, the patient will do better. There are 42 dyads enrolled in the study associated with caregivers that were randomized to the intervention.
- Health Information (Patient): The study also aims to explore the effect of caregiver outcomes on patient outcomes. The hypothesis is that if the caregiver is less stressed, the patient will do better. There are 51 dyads enrolled in the study associated with caregivers that were randomized to health information.
Arm/Group | Intervention | Health Information | Intervention (Patient) | Health Information (Patient)
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/125 | 15/42 | 12/51
Serious Adverse Events (participants affected / at risk) | 9/125 | 13/125 | 21/42 | 26/51
Other Adverse Events (participants affected / at risk) | 0/125 | 0/125 | 0/29 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=125) | Health Information (N=125) | Intervention (Patient) (N=42) | Health Information (Patient) (N=51)
COVID (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
RSV (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
allergy (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complications Due to Gall Stone Surgery (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COPD/Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Fall/fall complications (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 2 (2) | 4 (4)
gallbladder removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
gout (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
heart attack (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
high blood sugar (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
skin cancer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
stomach flu (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
stroke (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
vertigo (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 0 (0) | 12 (24) | 21 (34)
Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hemotology (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (7)
Immunology (Immune system disorders) | 0 (0) | 0 (0) | 6 (8) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Other (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations include enrollment from a single center although the center receives referrals from a diverse northeastern region of the US. Attrition was larger than anticipated and intervention engagement was variable. Although the sample enrolled was predominately White, female, and well-educated, it was large and diverse in many ways with almost 40% from groups who did not identify as White and almost 15% men.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT03988621/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT03988621/ICF_000.pdf